CLINICAL TRIAL: NCT05789186
Title: Clinical Study of Cang Ai Volatile Oil (CAVO) on Mild to Moderate Depression in Children and Adolescents
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chen Qian (Other)
Responsible Party: Sponsor-Investigator, Chen Qian, Yunnan University of Chinese Medicine, Yunnan University of Chinese Medicine
Organization: Yunnan University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAVO
Record Dates: First submitted 2023-02-11; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Depression
Keywords: Depression; Children; Adolescents; Aromatic Chinese Medicine
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test group (Experimental): CAVO aromatherapy patch at 3% concentration （continue sniffing for 15 minutes ）and Fluoxetine Hydrochloride mimetic （20mg/tablet，once a day，10mg each time）
  Interventions: Drug: CAVO aromatherapy patch at 3% concentration+Fluoxetine hydrochloride mimetic
- Positive drug group (Active Comparator): CAVO aromatherapy patch at 0.1% concentration（continue sniffing for 15 minutes ） and Fluoxetine hydrochloride tablet （20mg/tablet，once a day，10mg each time)
  Interventions: Drug: Fluoxetine hydrochloride tablet+CAVO aromatherapy patch at 0.1% concentration
- Blank control group (Sham Comparator): Concentration 0.1% CAVO aromatherapy patch（continue sniffing for 15 minutes）and fluoxetine hydrochloride mimetic（20mg/tablet，once a day，10mg each time）
  Interventions: Drug: Fluoxetine hydrochloride mimetic+CAVO aromatherapy patch at 0.1% concentration

INTERVENTIONS:
Drug: CAVO aromatherapy patch at 3% concentration+Fluoxetine hydrochloride mimetic — CAVO aromatherapy patch at 3% concentration enhances neuroelectrical activity in the brain (especially in the prefrontal cortex), exerting an antidepressant effect.Fluoxetine hydrochloride mimetic without drug treatment effect.
  Arms: Test group
Drug: Fluoxetine hydrochloride tablet+CAVO aromatherapy patch at 0.1% concentration — Fluoxetine hydrochloride tablet was widely used selective 5-HT reuptake inhibitor (SSRI) that selectively inhibits the 5-HT transporter, blocks the reuptake of 5-HT by the presynaptic membrane, and prolongs and increases the effects of 5-HT, resulting in antidepressant effects.CAVO aromatherapy patch at 0.1% concentration without drug treatment effect.
  Arms: Positive drug group
Drug: Fluoxetine hydrochloride mimetic+CAVO aromatherapy patch at 0.1% concentration — Placebo without drug treatment effect
  Arms: Blank control group

SUMMARY:
A randomized controlled trial was conducted to observe the improvement of mild to moderate depressive symptoms in children and adolescents with the aromatic herbal compound Cang Ai Volatile Oil (CAVO) and to evaluate the effectiveness and safety of the clinical application of CAVO.

DETAILED DESCRIPTION:
The trial was divided into: screening period, pre-treatment period, treatment period (first session, second session) and follow-up period.

(1) Screening period (14 days before intervention to 2 days before intervention): 108 patients with mild to moderate adolescent depression, regardless of gender, are to be enrolled. Patients will sign an informed consent form and will complete the screening period from the 14th pre-intervention day to the 2nd pre-intervention day.

(2) Pre-treatment (1 day prior to intervention): Patients who meet all inclusion criteria and do not meet any of the exclusion criteria will obtain a randomisation number 1 day prior to dosing and will be randomised in a 1:1:1 ratio to either the trial group (Group A), positive drug group (Group B) or blank control group (Group C). Subjects undergo an alcohol breath test and urine drug screen on an empty stomach at the test site to determine if they meet the entry criteria. Blood tests will be taken on an empty stomach on the day of the trial for testing, followed by food and 30 minutes later, blood pressure and EEG measurements will be taken and a depression scale will be completed after completion of NIR brain function measurements.

(3) Treatment period (first course: weeks 1 to 4, second course: weeks 5 to 8).

1. Test group: Each subject was given a sufficient amount of CAVO aromatherapy patch + fluoxetine hydrochloride mimetic at a concentration of 3%. The subject was instructed to fix the aromatherapy patch on the near-nasal part of the mouthpiece daily and complete two sniffing inhalations at fixed times (07:45-08:00 and 19:45-20:00) daily during the course of the treatment period, each time for 15 minutes, and to take 1 tablet of fluoxetine mimetic orally once a day. times.
2. Positive drug group: Each subject was given a sufficient amount of CAVO aromatherapy patch + fluoxetine hydrochloride tablet (20mg/tablet) at a concentration of 0.1%, and was instructed to take fluoxetine hydrochloride tablet (20mg/tablet) orally (10mg/dose, once a day). The aromatherapy patch was applied to the nasal area of the mask once a day.
3. Blank control group: Subjects were given a sufficient amount of CAVO aromatherapy patch + fluoxetine hydrochloride mimetic (20mg/tablet) at a concentration of 0.1% and were instructed to fix the aromatherapy patch on the near nasal area of the mouthpiece twice a day during the treatment period at fixed times (07:45-08:00 and 19:45-20:00) and to take 1 tablet of fluoxetine mimetic by mouth for 15 minutes each time. tablet of fluoxetine mimetic (20mg/tablet), 10mg/dose, once a day.

   Subjects will be required to complete blood pressure measurements, EEG measurements and NIR brain function measurements at the end of the first and second sessions respectively and then complete a depression rating scale. Blood will also need to be taken on an empty stomach at the end of the treatment period for submission for testing.
4. Follow-up period: (Week 9 to 10) Patients complete a follow-up examination at week 9 to 10 after the first dose. The investigator will continue to follow up with you by telephone for 1 week (at least 2 times, 1 day and 1 week after the end of the trial) to see how you are doing. You will be asked to answer a call back from your doctor and you will need to cooperate with the investigator's questioning.

ELIGIBILITY:
Inclusion Criteria:

* Meets the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and International Classification of Diseases (ICD) 10th Revision diagnostic criteria for mild to moderate depressive episodes, either first or recurrent, and not accompanied by psychotic symptoms.
* Meeting the diagnostic criteria for depression in Chinese medicine.
* 10 to 18 years of age (including borderline values), either sex.
* Depression scale: BDI-2, HAMD depression scale score of mild to moderate
* Healthy sense of smell, no allergic diseases or respiratory diseases.
* Have not used antidepressants and other psychiatric drugs or physiotherapy such as electroconvulsive or transcranial magnetic stimulation for at least 1 week prior to the examination.
* Depressive episodes lasting 2 weeks or more.
* All subjects have volunteered to participate and signed an informed consent form, as approved by the hospital's ethics committee.

Exclusion Criteria:

* A history of alcohol and drug dependence is strictly excluded.
* Current or prior diagnosis of a major psychiatric disorder other than depression consistent with DSM-5, such as bipolar disorder, neurodevelopmental disorder, neurocognitive disorder, schizophrenia, psychotic disorder, obsessive-compulsive disorder, panic disorder, post-traumatic stress disorder, antisocial personality disorder, etc.
* Depression with a history of organic brain disease and endocrine disorders or secondary to other psychiatric disorders.
* Persons at high risk of suicide: e.g., suicide attempts, recent suicide attempts, and those without family supervision
* Those with a history of manic or hypomanic episodes.
* Regularly taking antidepressants within 2 weeks prior to screening and not having discontinued psychotropic medication for 7 half-lives (at least 2 weeks for monoamine oxidase inhibitors and at least 1 month for fluoxetine) prior to randomisation to the group.
* Patients who have received physical therapy such as MECT, TMS, Vagus Nerve Stimulation (VNS), Deep Brain Stimulation (DBS), and other treatments such as light therapy, music therapy, exercise therapy, and acupuncture in the 3 months prior to screening.
* Patients with severe or unstable cardiovascular, respiratory, hepatic, renal, endocrine, haematological or other systemic disease which, in the opinion of the investigator, makes them unsuitable for enrollment in this study.
* Persons with known hypersensitivity to the test drug, or who are allergic.
* Those who have used the clinical trial drug within 3 months prior to the first dose, or those who plan to participate in other clinical trials during this study (ask, enquire).

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
The score of Hamilton Depression Scale(HAMD),Children's Depression Inventory(CDI). | 3 months
  The score of Hamilton Depression Scale(HAMD)>20，Total score 80 points，a total score of more than 35 on 24 items is considered severe depression, more than 20, possibly mild or moderate depression, and if less than 8, the patient has no depressive symptoms.
  The score of Children's Depression Inventory(CDI)>19，A scale of 0, 1 and 2 was used, indicating "occasionally", "often" and "always" respectively, indicating the frequency of symptoms, with a total score of 54. According to the original scale norm, 19 is the cut-off score for determining depressive symptoms, the higher the score the more severe the depression.
Serum pro-inflammatory cytokine assays, anti-inflammatory cytokines. | 3 months
  Serum pro-inflammatory cytokine assays include Tumour necrosis factor-alpha in pg/mg; Interleukin-1β in pg/mg; Interleukin-6 in pg/mg; Interferon gamma in pg/mg; Anti-inflammatory cytokines include Transforming growth factor-β in pg/mg; Interleukin-10 in pg/mg; Interleukin-4 in pg/mg; Interleukin-8 in pg/mg
HPA axis function test | 3 months
  Adrenocorticotropin-releasing hormone in μIU/ml； Pro-adrenocorticotropic hormone in μ IU/ml； Cortisol in μIU/ml
Serum glutamate, gamma-aminobutyric acid, 5-hydroxytryptamine levels. | 3 months
  Serum glutamate in μmol/L, Gamma-aminobutyric acid in μmol/L, 5-hydroxytryptamine in μmol/L

SECONDARY OUTCOMES:
Safety indicators Safety indicators | 3 months
  Heart rate in bpm,
Safety indicators Safety indicators | 3 months
  blood pressure include systolic and diastolic pressure in mmHg
Physical examination indicators（Liver function and kidney function） | 3 months
  Liver function include Alanine transaminase（ALT） in U/l; Aminotransferase aspartate（AST） in U/l;
Physical examination indicators（Liver function and kidney function） | 3 months
  Alkaline phosphatase（ALP） in G/L; Albumin（ALB） in G/L; Globulin(GLB) in G/L;
Physical examination indicators（Liver function and kidney function） | 3 months
  Total bilirubin（TBIL） in Umol/L;
Physical examination indicators（Liver function and kidney function） | 3 months
  Kidney function include Blood Urea Nitrogen（BUN）in mmol/L；
Physical examination indicators（Liver function and kidney function） | 3 months
  Creatinine(Cr）in μmol/（kg/d）.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Provincial Hospital of Traditional Chinese Medicine, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
References to deidentified individual participant data (IPD) sets and supporting information.